CLINICAL TRIAL: NCT05337475
Title: Feeding and Swallowing Problems in Infants With Laryngomalacia
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amal Fouad Sayed, Principal Investigator, Sohag University
Other Study IDs: Soh-Med-22-04-23
Record Dates: First submitted 2022-04-06; First posted 2022-04-20 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Feeding Disorders; Swallowing Disorder; Laryngomalacia
MeSH Terms: conditions — Feeding and Eating Disorders; Deglutition Disorders; Laryngomalacia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational cross-sectional study Infants with laryngomalacia Feeding and swallowing assessment

DETAILED DESCRIPTION:
Identification of swallowing and feeding disorders in infants with laryngomalacia.

Identify if there is relation between severity of laryngomalacia and feeding and swallowing disorder.

ELIGIBILITY:
Inclusion criteria:

* Infants up to 2 years old diagnosed with laryngomalacia.
* Full term infants.

Exclusion criteria:

* Infants with other possible causes of dysphagia e.g., craniofacial anomalies, BDMH and neurological affection secondary to birth trauma, hypoxic ischemic encephalopathy and other brain insults.
* Infants who were lethargic and/or medically unstable and were generally unable to participate to protocol of assessment.
* Premature infants.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with suspected laryngomalacia referred to phoniatrics unit, Sohag University Hospitals.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Mansoura Early Feeding Skills Assessment (MEFSA) | 2 years
  an 85-item observational measure of oral feeding skill. It will be used for assessing oral feeding through maturation of oral feeding skill. The MEFSA includes 3 main sections; pre-feeding, during feeding and post-feeding sections. The "during feeding" section, "Oral Feeding Maintenance" will be used in this study which supports infant based feeding that give the infant opportunity to communicate and express stress signals that must be respected. It proposed to observe the infant from moment to moment during feeding. This section composed of 30 items to assess infant abilities to (a) remain engaged in feeding, (b) organize oral-motor skills, (c) maintain physiologic stability and (d) coordinate SSB.
Fibreoptic Endoscopic Evaluation of swallowing (FEES) | 2 years
  FEES will be done with presentations of food and/or milk consistency (Secretions, thin and thick fluids, puree and/or solids) to obtain multiple trials of each texture. Infants who are fed only milk, FEES will be performed either with bottle-feeding or 5ml syringe (without needle) with the milk.
  Each infant will be fed by his or her typical caregiver or by the nurse. The feeding protocol began by presenting the infants with the bottle and/or nipple. If no aspiration occurred on the initial swallows, then the infant will be allowed to suck on the bottle until there was a change in swallowing function, 60 ml was finished, or the infant refused to suck.

SECONDARY OUTCOMES:
The Functional Oral Intake Scale- Suckle Feeds and Transitional Feeds (FOIS-SFTF) | 2 years
  score (1) stand for nothing by mouth, score (2) Tube dependent, with minimal attempts at liquids or food, score (3) Tube dependent, with consistent intake of liquids or food, score (4) Total oral diet, but requiring special preparation of liquids (ie, thickened liquids) +/- compensations, score (4.5) Total oral diet, but requiring special preparation of solids (eg, foods of different texture and/or liquid supplements) +/- compensations, score (5) Total oral diet, without special preparation (ie, regular thin fluids, foods of same texture as peers, and no additional liquid supplements), but with compensations, score (6) Total oral diet, with no restrictions

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospitals, Sohag, Sohag Governorate, Egypt